CLINICAL TRIAL: NCT01537809
Title: The Impact of Vitamin D Supplementation on Cardiometabolic Risk Factors in Schoolchildren
Brief Title: Impact of Vitamin D Supplementation on Cardiometabolic Risk Factors [The Daily D Health Study]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Office of Dietary Supplements (ODS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston University (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1103016; 3R01HL106160 (NIH)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Vitamin D Deficiency; Avitaminosis; Deficiency Diseases; Blood lipids
MeSH Terms: conditions — Vitamin D Deficiency; Avitaminosis; Deficiency Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- D3 600 IU/ daily (Active Comparator): Subjects randomized to 600 IU/day of vitamin D3 taken orally for six months.
  Interventions: Dietary Supplement: Vitamin D3
- D3 1000 IU/ daily (Active Comparator): Subjects randomized to 1000 IU/day of vitamin D3 taken orally for six months.
  Interventions: Dietary Supplement: Vitamin D3
- D3: 2000 IU/daily (Active Comparator): Subjects randomized to 2000 IU/day of vitamin D3 taken orally for six months.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Subjects are told to take vitamin D daily for 6 months.
Dietary Supplement: Vitamin D3 — Subjects are asked to take vitamin D orally, daily for six months.

SUMMARY:
The purpose of this research is to determine what supplemental doses of vitamin D may be necessary to raise serum levels to optimal levels and how vitamin D supplementation and changes in vitamin D status impact cardiovascular risk factors in schoolchildren.

DETAILED DESCRIPTION:
Research suggests that vitamin D, known mainly for its role in bone health, may have other roles in the body and that vitamin D deficiency may contribute to certain chronic diseases, such as cardiovascular disease. Recently, vitamin D has received growing attention due to the increased awareness of possible deficiencies among certain populations at risk of vitamin D deficiency. Most circulating 25-hydroxyvitamin D comes from exposure to UVB rays in natural sunlight. In 2010, the Institute of Medicine issued new recommendations that daily vitamin D intakes should be increased to 600 IU/day for children ages 1-18. However, even with these recommendations in place, roughly 20% of all children are below the recommended 20 ng/mL. Moreover, more than two-thirds of all children have levels below 30 ng/mL, including 80% of Hispanic children and 92% of non-Hispanic black children. Therefore, it is imperative to gain an understanding of: 1) what supplemental doses may be necessary for schoolchildren who are already at a disadvantage in achieving optimal levels of 25(OH)D due to factors such as living at a northern latitude, having high obesity rates, and where a large proportion of the population are Latino or African American; and 2) whether serum concentrations of 25(OH)D over 30 ng/mL in children prevent health risks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in 4th-8th grade
* Subjects must attend school where study is being conducted
* Subject and parent/guardian must give assent/consent to participate in study Related Requirements
* Subjects must complete all study visits (baseline, 3,6 and 12 months)
* Subjects must agree to be blinded

Exclusion Criteria:

* Subjects taking glucocorticoids
* Subjects not in 4th-8th grade
* Clinical diagnosis of Cystic Fibrosis
* Clinical diagnosis of Kidney disease
* Subjects currently taking a vitamin D supplement of >1000 IU/day
* Subjects diagnosed with Irritable Bowel Syndrome (IBS)
* Clinical diagnosis of AIDS
* Clinical diagnosis of Sarcoidosis
* Clinical diagnosis of Epilepsy

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 691 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D levels over six month period | Six months
  Subjects will be randomized to receive one of three doses of vitamin D3. Baseline serum 25(OH)D levels will be compared to serum 25(OH)D at 3 and 6 months.
  Safety Issue?: (FDAAA) No

SECONDARY OUTCOMES:
measure serum glucose and blood lipids (total cholesterol, HDL, LDL and triglycerides) in connection with changes in vitamin D status | 12 months
  Baseline cardiometabolic risk factors will be compared at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sacheck, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sacheck J, Goodman E, Chui K, Chomitz V, Must A, Economos C. Vitamin D deficiency, adiposity, and cardiometabolic risk in urban schoolchildren. J Pediatr. 2011 Dec;159(6):945-50. doi: 10.1016/j.jpeds.2011.06.001. Epub 2011 Jul 23. PMID 21784451
- [Derived] Sacheck JM, Huang Q, Van Rompay MI, Chomitz VR, Economos CD, Eliasziw M, Gordon CM, Goodman E. Vitamin D supplementation and cardiometabolic risk factors among diverse schoolchildren: a randomized clinical trial. Am J Clin Nutr. 2022 Jan 11;115(1):73-82. doi: 10.1093/ajcn/nqab319. PMID 34550329
- [Derived] Blakeley CE, Van Rompay MI, Schultz NS, Sacheck JM. Relationship between muscle strength and dyslipidemia, serum 25(OH)D, and weight status among diverse schoolchildren: a cross-sectional analysis. BMC Pediatr. 2018 Feb 2;18(1):23. doi: 10.1186/s12887-018-0998-x. PMID 29394922
- [Derived] Sacheck JM, Van Rompay MI, Chomitz VR, Economos CD, Eliasziw M, Goodman E, Gordon CM, Holick MF. Impact of Three Doses of Vitamin D3 on Serum 25(OH)D Deficiency and Insufficiency in At-Risk Schoolchildren. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4496-4505. doi: 10.1210/jc.2017-01179. PMID 29029097
- [Derived] Sawicki CM, Van Rompay MI, Au LE, Gordon CM, Sacheck JM. Sun-Exposed Skin Color Is Associated with Changes in Serum 25-Hydroxyvitamin D in Racially/Ethnically Diverse Children. J Nutr. 2016 Apr;146(4):751-7. doi: 10.3945/jn.115.222505. Epub 2016 Mar 2. PMID 26936138
- [Derived] Van Rompay MI, McKeown NM, Goodman E, Eliasziw M, Chomitz VR, Gordon CM, Economos CD, Sacheck JM. Sugar-Sweetened Beverage Intake Is Positively Associated with Baseline Triglyceride Concentrations, and Changes in Intake Are Inversely Associated with Changes in HDL Cholesterol over 12 Months in a Multi-Ethnic Sample of Children. J Nutr. 2015 Oct;145(10):2389-95. doi: 10.3945/jn.115.212662. Epub 2015 Sep 2. PMID 26338888